CLINICAL TRIAL: NCT02956486
Title: A Placebo-Controlled, Double-Blind, Parallel-Group, 24 Month Study With an Open-Label Extension Phase to Evaluate the Efficacy and Safety of Elenbecestat (E2609) in Subjects With Early Alzheimer's Disease
Brief Title: A 24-Month Study to Evaluate the Efficacy and Safety of Elenbecestat (E2609) in Participants With Early Alzheimer's Disease
Acronym: MissionAD1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to an unfavorable risk-benefit ratio including no evidence of potential efficacy, and the adverse event profile of E2609 being worse than placebo.
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2609-G000-301; 2016-003928-23 (EudraCT Number); 2016-004128-42 (EudraCT Number); NCT03036280 (obsolete NCT alias)
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer's Disease
Keywords: Elenbecestat; E2609; Alzheimer's Disease; Early Alzheimer's Disease; Prodromal Alzheimer's Disease; Dementia; Dementia, Alzheimer's type; Mild Cognitive Impairment; MissionAD1
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Core Study: Elenbecestat 50 mg (Experimental): Participants will receive one 50 milligram (mg) elenbecestat tablet, orally, once a day in the morning. The core study will be double blinded.
  Interventions: Drug: Elenbecestat
- Core Study: Placebo (Placebo Comparator): Participants will receive one matching placebo tablet, orally, once a day in the morning. The core study will be double blinded.
  Interventions: Drug: Placebo
- Open-label Extension Phase: Elenbecestat 50 mg (Experimental): Participants completing the core study will receive one 50 mg elenbecestat tablet, orally, once a day in the morning.
  Interventions: Drug: Elenbecestat

INTERVENTIONS:
Drug: Elenbecestat — Oral tablet.
  Other Names: E2609
  Arms: Core Study: Elenbecestat 50 mg; Open-label Extension Phase: Elenbecestat 50 mg
Drug: Placebo — Oral tablet.
  Arms: Core Study: Placebo

SUMMARY:
The name of this trial is MissionAD1. This phase 3 study consists of a Core and Open Label Extension (OLE) Phase in participants with Early Alzheimer's Disease (EAD), and will be conducted to evaluate the efficacy and safety of E2609. The Core is a 24-month treatment, multicenter, double blind, placebo controlled parallel group study. The OLE is a 24-month treatment, one group study. The data for the studies E2609-G000-301 (NCT02956486, MissionAD1) and E2609-G000-302 (NCT03036280, MissionAD2) will be pooled.

ELIGIBILITY:
Inclusion Criteria:

Core Study

* Mild cognitive impairment due to Alzheimer's disease (AD) or mild AD dementia including

  1. Mini Mental State Examination score equal to or greater than 24
  2. Clinical Dementia Rating (CDR) global score of 0.5
  3. CDR Memory Box score of 0.5 or greater
* Impaired episodic memory confirmed by a list learning task
* Positive biomarker for brain amyloid pathology as indicated by either amyloid positron emission tomography or cerebrospinal fluid AD assessment or both

Extension Phase

• Participants who complete the Core Study

Exclusion Criteria:

Core Study

* Females who are breastfeeding or pregnant at Screening or Baseline. Females of child-bearing potential must use a highly effective method of contraception throughout the entire study period and for 28 days after study drug discontinuation
* Any condition that may be contributing to cognitive impairment above and beyond that caused by the participant's AD
* Participants with a history of seizures within 5 years of Screening
* History of transient ischemic attacks or stroke within 12 months of Screening
* Psychiatric diagnosis or symptoms (example, hallucinations, major depression, delusions etc.)
* Suicidal ideation or any suicidal behavior within 6 months before Screening or has been hospitalized or treated for suicidal behavior in the past 5 years
* Have any contraindications to magnetic resonance imaging (MRI) scanning or

  1. Have lesions that could indicate a dementia diagnosis other than AD on brain MRI
  2. Exhibit other significant pathological findings on brain MRI.
* Participants who have a history of moderate to severe hepatic impairment (example, Child-Pugh Class B or C)
* Results of laboratory tests conducted during Screening that are outside the following limits:

  1. Absolute lymphocyte count below the lower limit of normal (LLN)
  2. Thyroid stimulating hormone above normal range
  3. Abnormally low Vitamin B12 levels
* Participants at increased risk of infection
* Have received any live vaccine/live attenuated vaccine in the 3 months before randomization
* Any chronic inflammatory disease that is not adequately controlled or that requires systemic immunosuppressive or immunomodulatory therapy
* Any other clinically significant abnormalities
* Severe visual or hearing impairment
* A prolonged corrected QT (QTc) interval (QT interval with Fridericia's correction [QTcF] greater than 450 milliseconds [ms])
* Malignant neoplasms within 5 years of Screening
* Known or suspected history of drug or alcohol abuse
* Taking prohibited medications, which must be reviewed with the Investigator
* Have participated in a recent clinical study

Note: Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2212 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (258):
- United States (88):
  - Facility #1, Chandler, Arizona
  - Facility #1, Colton, California
  - Facility #1, Costa Mesa, California
  - Facility #1, Fullerton, California
  - Facility #1, Imperial, California
  - Facility #1, Irvine, California
  - Facility #1, Lemon Grove, California
  - Facility #1, Oceanside, California
  - Facility #2, Oceanside, California
  - Facility #1, Oxnard, California
  - Facility #1, Panorama City, California
  - Facility #1, San Diego, California
  - Facility #1, Denver, Colorado
  - Facility #1, Atlantis, Florida
  - Facility #1, Aventura, Florida
  - Facility #2, Aventura, Florida
  - Facility #1, Boynton Beach, Florida
  - Facility #1, Coral Gables, Florida
  - Facility #2, Coral Gables, Florida
  - Facility #1, Delray Beach, Florida
  - Facility #1, Doral, Florida
  - Facility #1, Hialeah, Florida
  - Facility #2, Miami, Florida
  - Facility #11, Miami, Florida
  - Facility #9, Miami, Florida
  - Facility #10, Miami, Florida
  - Facility #4, Miami, Florida
  - Facility #1, Miami, Florida
  - Facility #6, Miami, Florida
  - Facility #3, Miami, Florida
  - Facility #7, Miami, Florida
  - Facility #8, Miami, Florida
  - Facility #2, Orlando, Florida
  - Facility #1, Orlando, Florida
  - Facility #3, Orlando, Florida
  - Facility #1, Palm Beach Gardens, Florida
  - Facility #1, Pompano Beach, Florida
  - Facility #1, Port Charlotte, Florida
  - Facility #1, Port Orange, Florida
  - Facility #1, Spring Hill, Florida
  - Facility #1, Tampa, Florida
  - Facility #2, Tampa, Florida
  - Facility #1, The Villages, Florida
  - Facility #1, Atlanta, Georgia
  - Facility #1, Columbus, Georgia
  - Facility #1, Decatur, Georgia
  - Facility #1, Suwanee, Georgia
  - Facility #1, Meridian, Idaho
  - Facility #1, Northbrook, Illinois
  - Facility #2, Wichita, Kansas
  - Facility #1, Boston, Massachusetts
  - Facility #1, Farmington Hills, Michigan
  - Facility #1, Chesterfield, Missouri
  - Facility #1, City of Saint Peters, Missouri
  - Facility #1, O'Fallon, Missouri
  - Facility #2, St Louis, Missouri
  - Facility #1, Mount Arlington, New Jersey
  - Facility #2, Springfield, New Jersey
  - Facility #1, West Long Branch, New Jersey
  - Facility #1, Amherst, New York
  - Facility #1, Brooklyn, New York
  - Facility #1, New York, New York
  - Facility #1, Canton, Ohio
  - Facility #1, Centerville, Ohio
  - Facility #1, Cleveland, Ohio
  - Facility #1, Dayton, Ohio
  - Facility #1, Lakewood, Ohio
  - Facility #1, Westerville, Ohio
  - Facility #1, Oklahoma City, Oklahoma
  - Facility #1, Portland, Oregon
  - Facility #1, Jenkintown, Pennsylvania
  - Facility #1, Media, Pennsylvania
  - Facility #1, Philadelphia, Pennsylvania
  - Facility #1, East Providence, Rhode Island
  - Facility #1, Providence, Rhode Island
  - Facility #1, Port Royal, South Carolina
  - Facility #1, Cordova, Tennessee
  - Facility #2, Nashville, Tennessee
  - Facility #1, Nashville, Tennessee
  - Facility #1, Austin, Texas
  - Facility #1, Dallas, Texas
  - Facility #1, Houston, Texas
  - Facility #1, San Antonio, Texas
  - Facility #3, San Antonio, Texas
  - Facility #1, Salt Lake City, Utah
  - Facility #1, Bennington, Vermont
  - Facility #1, Hampton, Virginia
  - Facility #1, Madison, Wisconsin
- Argentina (14):
  - Facility #2, Caba, Buenos Aires
  - Facility #1, Caba, Buenos Aires
  - Facility #4, Caba, Buenos Aires
  - Facility #3, Caba, Buenos Aires
  - Facility #1, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Facility #3, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Facility #2, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Facility #1, Córdoba, Capital
  - Facility #1, Rosario, Santa Fe Province
  - Facility #4, Buenos Aires
  - Facility #5, Caba
  - Facility #2, Córdoba
  - Facility #3, Córdoba
  - Facility #1, Santa Fe
- Australia (12):
  - Facility #1, Darlinghurst, New South Wales
  - Facility #1, Macquarie Park, New South Wales
  - Facility #1, Tumbi Vmbi, New South Wales
  - Facility #1, Brisbane, Queensland
  - Facility #1, Caulfield, Victoria
  - Facility #1, Geelong, Victoria
  - Facility #1, Heidelberg, Victoria
  - Facility #1, Malvern, Victoria
  - Facility #2, Melbourne, Victoria
  - Facility #1, Parkville, Victoria
  - Facility #1, Nedlands, Western Australia
  - Facility #3, Melbourne
- Facility #1, Vienna, Austria
- Bulgaria (7):
  - Facility #1, Pleven
  - Facility #1, Plovdiv
  - Facility #1, Rousse
  - Facility #4, Sofia
  - Facility #3, Sofia
  - Facility #1, Sofia
  - Facility #2, Sofia
- Canada (9):
  - Facility #1, Kamloops, British Columbia
  - Facility #1, Kelowna, British Columbia
  - Facility #1, West Vancouver, British Columbia
  - Facility #1, Halifax, Nova Scotia
  - Facility #1, Kentville, Nova Scotia
  - Facility #1, Ottawa, Ontario
  - Facility #1, Peterborough, Ontario
  - Facility #1, Montreal, Quebec
  - Facility #1, Sherbrooke, Quebec
- Czechia (4):
  - Facility #1, Hradec Králové
  - Facility #1, Kladno
  - Facility #1, Olomouc
  - Facility #1, Prague
- France (8):
  - Facility #1, Montpellier, Herault
  - Facility #1, Bordeaux
  - Facility #1, Bron
  - Facility #1, Marseille
  - Facility #1, Nantes
  - Facility #1, Paris
  - Facility #1, Rouen
  - Facility #1, Toulouse
- Germany (10):
  - Facility #1, Neuburg am Inn, Bavaria
  - Facility #1, Hoppegarten, Brandenburg
  - Facility #1, Oranienburg, Brandenburg
  - Facility #1, Frankfurt am Main, Hesse
  - Facility #1, Leipzig, Saxony
  - Facility #1, Berlin
  - Facility #2, Berlin
  - Facility #1, Gera
  - Facility #1, Homburg/Saar
  - Facility #1, Schwerin
- Greece (2):
  - Facility #5, Athens
  - Facility #4, Athens
- Japan (48):
  - Eisai Trial Site 1, Anjo-shi, Aichi-ken
  - Eisai Trial Site 1, Nagoya, Aichi-ken
  - Eisai Trial Site 1, Obu-shi, Aichi-ken
  - Eisai Trial Site 1, Yoshida-gun, Fukui
  - Eisai Trail Site 1, Kitakyushu-shi, Fukuoka
  - Eisai Trial Site 1, Omuta-shi, Fukuoka
  - Eisai Trial Site 1, Fujioka-shi, Gunma
  - Eisai Trial Site 1, Otake-shi, Hiroshima
  - Eisai Trial Site 1, Himeji, Hyōgo
  - Eisai Trial Site 2, Himeji-shi, Hyōgo
  - Eisai Trial Site 1, Kobe, Hyōgo
  - Facility #1, Hiragi, Kagawa-ken
  - Eisai Trial Site 3, Takamatsu, Kagawa-ken
  - Eisai Trial Site 1, Fujisawa-shi, Kanagawa
  - Eisai Trial Site 1, Kyoto, Kyoto
  - Eisai Trial Site 2, Kyoto, Kyoto
  - Eisai Trial site 5, Kyoto, Kyoto
  - Eisai Trial Site 4, Kyoto, Kyoto
  - Eisai Trial Site 1, Shimogyo-ku, Kyoto
  - Eisai Trial Site 1, Higashimorokatagun, Miyazaki
  - Eisai Trial Site 1, Kurashiki-shi, Okayama-ken
  - Eisai Trial Site 2, Kurashiki-shi, Okayama-ken
  - Eisai Trial Site 1, Okayama, Okayama-ken
  - Eisai Trial Site 2, Okayama, Okayama-ken
  - Eisai Trial Site 1, Hirakata, Osaka
  - Eisai Trial Site 1, Naniwa-Ku, Osaka
  - Eisai Trial Site 1, Osaka, Osaka
  - Eisai Trial Site 3, Osaka, Osaka
  - Eisai Trial Site 2, Osaka, Osaka
  - Eisai Trial site 2, Sakai-shi, Osaka
  - Eisai Trial Site 1, Suita-shi, Osaka
  - Eisai Trial Site 2, Suita-shi, Osaka
  - Eisai Trial Site 1, Suminoe-ku, Osaka
  - Eisai Trial Site 1, Kanzaki-gun, Saga-ken
  - Eisai Trial Site 2, Ōtsu, Shiga
  - Eisai Trial Site 1, Ōtsu, Shiga
  - Eisai Trial Site 1, Tokushima, Tokushima
  - Eisai Trial Site 1, Bunkyo-ku, Tokyo
  - Eisai Trial Site 2, Bunkyo-ku, Tokyo
  - Eisai Trial Site 1, Kodaira-shi, Tokyo
  - Eisai Trial Site 1, Minato-ku, Tokyo
  - Eisai Trial Site 1, Setagaya-ku, Tokyo
  - Eisai Trial Site 1, Shinjuku-ku, Tokyo
  - Eisai Trial Site 1, Sumida-ku, Tokyo
  - Eisai Trial Site 1, Hofu-shi, Yamaguchi
  - Eisai Trial Site 1, Kumamoto
  - Eisai Trial Site 3, Kyoto
  - Eisai Trial Site 1, Osaka
- Poland (7):
  - Facility #1, Katowice
  - Facility #1, Kielce
  - Facility #1, Krakow
  - Facility #1, Poznan
  - Facility #1, Poznari
  - Facility #1, Siemianowice Śląskie
  - Facility #1, Warsaw
- Facility #1, Guimarães, Portugal
- Facility #1, Moscow, Russia
- Facility #1, Bratislava, Slovakia
- South Korea (10):
  - Facility #1, Bucheon-si, Gyeonggi-do
  - Facility #1, Seongnam-si, Gyeonggi-do
  - Facility #1, Busan
  - Facility #1, Incheon
  - Facility #5, Seoul
  - Facility #3, Seoul
  - Facility #1, Seoul
  - Facility #4, Seoul
  - Facility #6, Seoul
  - Facility #2, Seoul
- Spain (11):
  - Facility #1, Elche, Alicante
  - Facility #1, Palma de Mallorca, Balearic Islands
  - Facility #1, Sant Cugat del Vallès, Barcelona
  - Facility #1, Getxo, Bizkaia
  - Facility #1, Donostia / San Sebastian, Gipuzkoa
  - Facility #1, El Palmar, Murcia
  - Facility #1, Barcelona
  - Facility #2, Madrid
  - Facility #1, Madrid
  - Facility #1, Valencia
  - Facility #2, Valencia
- United Kingdom (24):
  - Facility #1, Cambridge, Cambridgeshire
  - Facility #1, Chester, Cheshire
  - Facility #1, Winwick, Warrington, Cheshire
  - Facility #1, Plymouth, Devon
  - Facility #1, Bournemouth, Dorset
  - Facility #1, Crowborough, East Sussex
  - Facility #1, Manchester, Greater Manchester
  - Facility #1, Southampton, Hampshire
  - Facility #1, Glasgow, Lanarkshire
  - Facility #1, Blackpool, Lancashire
  - Facility #1, Preston, Lancashire
  - Facility #2, London, Middlesex
  - Facility #1, Bath, North East Somerset
  - Facility #1, Oxford, Oxfordshire
  - Facility #1, Aberdeen, Scotland
  - Facility #1, Sheffield, South Yorkshire
  - Facility #1, Leatherhead, Surrey
  - Facility #1, Birmingham, West Midlands
  - Facility #1, Swindon, Wilts
  - Facility #2, Glasgow
  - Facility #1, Guildford
  - Facility #1, London
  - Facility #4, London
  - Facility #3, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Devanarayan V, Doherty T, Charil A, Sachdev P, Ye Y, Murali LK, Llano DA, Zhou J, Reyderman L, Hampel H, Kramer LD, Dhadda S, Irizarry MC. Plasma pTau217 predicts continuous brain amyloid levels in preclinical and early Alzheimer's disease. Alzheimers Dement. 2024 Aug;20(8):5617-5628. doi: 10.1002/alz.14073. Epub 2024 Jun 28. PMID 38940656
- [Derived] Devanarayan V, Ye Y, Charil A, Andreozzi E, Sachdev P, Llano DA, Tian L, Zhu L, Hampel H, Kramer L, Dhadda S, Irizarry M; Alzheimer's Disease Neuroimaging Initiative (ADNI). Predicting clinical progression trajectories of early Alzheimer's disease patients. Alzheimers Dement. 2024 Mar;20(3):1725-1738. doi: 10.1002/alz.13565. Epub 2023 Dec 13. PMID 38087949
- [Derived] Bullich S, Mueller A, De Santi S, Koglin N, Krause S, Kaplow J, Kanekiyo M, Roe-Vellve N, Perrotin A, Jovalekic A, Scott D, Gee M, Stephens A, Irizarry M. Evaluation of tau deposition using 18F-PI-2620 PET in MCI and early AD subjects-a MissionAD tau sub-study. Alzheimers Res Ther. 2022 Jul 27;14(1):105. doi: 10.1186/s13195-022-01048-x. PMID 35897078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 426 investigative sites in China, Bulgaria, Croatia, Czech Republic, Greece, Hungary, Poland, Russia, Slovakia, Japan, Canada, Singapore, South Korea, Taiwan, Argentina, Chile, Mexico, Australia, Austria, Denmark, Finland, France, Germany, Italy, Portugal, South Africa, Spain, United Kingdom and the United States from 20 October 2016 to 15 January 2020.
Pre-assignment Details: This study included 2 parts: Core Phase and Extension Phase. A total of 9758 participants were screened, of which 7546 participants were screen failures and 2212 participants were randomized in the study. The data for the studies E2609-G000-301 (NCT02956486, MissionAD1) and E2609-G000-302 (NCT03036280, MissionAD2) was pooled.
Groups:
- Core Phase: Placebo: Participants received one elenbecestat matching-placebo tablet, orally, once daily in the morning with or without food up to 24 months. Participants were followed up for 3 months after last dose of elenbecestat matched placebo in core phase.
- Core Phase: Elenbecestat 50 mg: Participants received one elenbecestat 50 milligram (mg) tablet, orally, once daily in the morning with or without food up to 24 months. Participants were followed up for 3 months after last dose of elenbecestat in core phase.
- Extension Phase: Elenbecestat 50 mg: Eligible participants who completed the core phase entered the extension phase and received one elenbecestat 50 mg tablet, orally, once daily in the morning with or without food until commercial availability of elenbecestat, or a lack of positive benefit-risk assessment was determined, whichever occurred first. Participants were followed up for 1 month after the last dose of elenbecestat in the extension phase.
Period: Core Phase
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg | Extension Phase: Elenbecestat 50 mg
Started | 1108 | 1104 | 0
Treated | 1108 | 1101 | 0
Safety Analysis Set (SAS) | 1105 | 1099 | 0
Full Analysis Set (FAS) | 1084 | 1062 | 0
Completed | 29 | 32 | 0
Not Completed | 1079 | 1072 | 0
Not completed — Adverse Event | 51 | 88 | 0
Not completed — Lost to Follow-up | 8 | 6 | 0
Not completed — Inadequate therapeutic effect | 4 | 5 | 0
Not completed — Withdrawal by Subject | 101 | 104 | 0
Not completed — Study terminated by sponsor | 888 | 848 | 0
Not completed — Other | 27 | 18 | 0
Not completed — Not treated | 0 | 3 | 0
Period: Extension Phase
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg | Extension Phase: Elenbecestat 50 mg
Started | 0 | 0 | 19 (Eligible participants who completed core and consented for extension phase, entered extension phase.)
Treated | 0 | 0 | 18
Safety Analysis Set (SAS) | 0 | 0 | 18
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 19
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 16
Not completed — Not Treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The SAS was the group of participants who received at least 1 dose of study drug in the core phase and had at least 1 post-dose safety assessment.
Groups:
- Core Phase: Elenbecestat 50 mg: Participants received one elenbecestat 50 mg tablet, orally, once daily in the morning with or without food up to 24 months. Participants were followed up for 3 months after last dose of elenbecestat in core phase.
- Total: Total of all reporting groups
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg | Total
Number analyzed (Participants) | 1105 | 1099 | 2204
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (7.09) | 71.9 (7.18) | 72.0 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 592 | 534 | 1126
  Male | 513 | 565 | 1078
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 162 | 158 | 320
  Not Hispanic or Latino | 943 | 941 | 1884
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 233 | 247 | 480
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 12 | 22 | 34
  White | 851 | 817 | 1668
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Change From Baseline up to Month 24 in the Clinical Dementia Rating-sum of Boxes (CDR-SB) Score
Description: The clinical dementia rating (CDR) scale is a clinical global rating scale that requires interviewing both the participant and an informant who knows and has contact with the participant. The CDR scale is a clinician directed assessment of both cognition and function, and is intended to capture the state and therefore the disease stage of the participant. The CDR scale assesses 6 domains of participant function (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment=0, questionable impairment=0.5, mild impairment=1, moderate impairment=2 and severe impairment=3. The CDR-SB is a sum of the individual domain scores and ranges from 0 to 18. Higher score indicates more impairment.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug in the core phase and had baseline and at least 1 post-dose primary efficacy measurement. Here "overall number of participants analyzed" signifies all participants included in mixed effects model for repeated measures (MMRM) who were evaluable for this specific outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1078 | 1053
score on a scale | 2.17 (0.142) | 1.99 (0.146)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; Analysis was based on the MMRM and factors for treatment group, visit, treatment group by visit interaction, clinical disease staging (mild cognitive impairment [MCI]/Prodromal, mild alzheimer's disease [AD]), concurrent AD medication use, region, apolipoprotein E (ApoE4) status (positive, negative) as fixed effects, and the baseline value and the baseline value by visit interaction as covariate; Test type: Superiority; p = 0.385, MMRM; Least Square (LS) Mean Difference = -0.17, 95% CI 2-sided [-0.57 to 0.22]

2. Primary Outcome: Extension Phase: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an adverse event that emerged during treatment or within 28 days following the last dose of study drug, having been absent at pretreatment (Baseline) or reemerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the adverse event was continuous. Number of participants with TEAEs (serious and non-serious adverse events) were reported based on their safety assessments of laboratory tests, suicidal ideation and suicidal behavior, drug abuse potential, physical examination, neurological examination, regular measurement of vital signs, magnetic resonance imaging and electrocardiogram parameter values.
Time Frame: From first dose of study drug up to approximately 6 months (including 1 month follow up) for the extension phase
Population: All safety participants was the group of participants who enrolled into the extension phase and received at least 1 dose of study drug in the extension phase.
Measure: Count of Participants; unit: Participants
Groups:
- Extension Phase: Elenbecestat 50 mg: In the extension phase, participants received one elenbecestat 50 mg tablet, orally, once daily in the morning with or without food until commercial availability of elenbecestat, or a lack of positive benefit-risk assessment was determined, whichever occurred first. Participants were followed up for 1 month after the last dose of elenbecestat in the extension phase.
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 18
Participants | 6

3. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in Alzheimer's Disease Composite Score (ADCOMS)
Description: ADCOMS is a weighted linear combination of 12 items from three existing clinical scales: the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog), the Mini Mental State Examination (MMSE), and the CDR. Four items are from the ADAS-cog (A4 [Delayed Word Recall], A7 [Orientation], A8 [Word Recognition], A11 [Word Finding]); 2 items are from the MMSE (M1 [Orientation Time], M7 [Drawing]); 6 items are from the CDR (C1 [Personal Care], C2 [Community Affairs], C3 [Home and Hobbies], C4 [Judgment and Problem Solving], C5 [Memory], C6 [Orientation]). Composite score is derived from the variables from the 12 items, and ranges from 0 to 1.97, where higher score indicates worse performance.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug in the core phase and had baseline and at least 1 post-dose primary efficacy measurement. Here "overall number of participants analyzed" signifies all participants included in MMRM who were evaluable for this specific outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1018 | 981
score on a scale | 0.24 (0.014) | 0.23 (0.015)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; Analysis was based on the MMRM and factors for treatment group, visit, treatment group by visit interaction, clinical disease staging (MCI/Prodromal, mild AD), concurrent AD medication use, region, ApoE4 status (positive, negative) as fixed effects, and the baseline value and the baseline value by visit interaction as covariate; Test type: Superiority; p = 0.345, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.06 to 0.02]

4. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in Amyloid Positron Emission Tomography (PET) Standardized Uptake Value Ratio (SUVR)
Description: Amyloid PET scan assesses cerebral amyloid load using 3 tracers (florbetapir, florbetaben and flutemetamol) which is standardized into centiloids for evaluation of AD. Centiloid values on centiloid scale is based on mean composite SUVR in cingulate, frontal, parietal and temporal cortexes using whole cerebellum as reference region. SUVR is ratio of tracer uptake in each of cingulate, frontal, parietal and temporal cortexes relative to cerebellum. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scans.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: The pharmacodynamic (PD) analysis set was the group of participants in the core phase who had sufficient PD data to derive at least 1 PD parameter. Here "overall number of participants analyzed" signifies all participants included in MMRM who were evaluable for this specific outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 268 | 248
score on a scale | 7.81 (2.500) | -5.02 (2.046)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < .001, MMRM; LS Mean Difference = -12.83, 95% CI 2-sided [-18.79 to -6.88]

5. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the CDR-SB Score for Participants Enriched by Baseline Amyloid PET SUVR Between 1.2 and 1.6
Description: The CDR scale is a clinical global rating scale that requires interviewing both the participant and an informant who knows and has contact with the participant. The CDR scale is a clinician directed assessment of both cognition and function, and is intended to capture the state and therefore the disease stage of the participant. The CDR scale assesses 6 domains of participant function (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment=0, questionable impairment=0.5, mild impairment=1, moderate impairment=2 and severe impairment=3. The CDR-SB is a sum of the individual domain scores and ranges from 0 to 18. Higher score indicates more impairment. Amyloid PET scans allow in vivo assessment of cerebral amyloid load. SUVR indicates the ratio of tracer uptake in the frontal cortex relative to the cerebellum or the ratio of tracer uptake in the whole brain relative to the cerebellum.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 664 | 617
score on a scale | 1.97 (0.157) | 1.74 (0.169)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.316, MMRM; LS Mean Difference = -0.23, 95% CI 2-sided [-0.67 to 0.22]

6. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the ADCOMS for Participants Enriched by Baseline Amyloid PET SUVR Between 1.2 and 1.6
Description: ADCOMS is a weighted linear combination of 12 items from three existing clinical scales: the ADAS-cog, the MMSE, and the CDR. Four items are from the ADAS-cog (A4 [Delayed Word Recall], A7 [Orientation], A8 [Word Recognition], A11 [Word Finding]); 2 items are from the MMSE (M1 [Orientation Time], M7 [Drawing]); 6 items are from the CDR (C1 [Personal Care], C2 [Community Affairs], C3 [Home and Hobbies], C4 [Judgment and Problem Solving], C5 [Memory], C6 [Orientation]). Composite score is derived from the variables from the 12 items, and ranges from 0 to 1.97, where higher score indicates worse performance. Amyloid PET scans allow in vivo assessment of cerebral amyloid load. SUVR indicates the ratio of tracer uptake in the frontal cortex relative to the cerebellum or the ratio of tracer uptake in the whole brain relative to the cerebellum.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 627 | 571
score on a scale | 0.23 (0.017) | 0.20 (0.018)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.254, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.07 to 0.02]

7. Secondary Outcome: Core Phase: Change Per Year (Mean Slope) in CDR-SB Score up to Month 24
Description: The CDR scale is a clinical global rating scale that requires interviewing both the participant and an informant who knows and has contact with the participant. The CDR scale is a clinician directed assessment of both cognition and function, and is intended to capture the state and therefore the disease stage of the participant. The CDR scale assesses 6 domains of participant function (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment=0, questionable impairment=0.5, mild impairment=1, moderate impairment=2 and severe impairment=3. The CDR-SB is a sum of the individual domain scores and ranges from 0 to 18. Higher score indicates more impairment. In this outcome measure, change per year (mean slope) in CDR-SB score was calculated up to month 24, where higher change indicated more impairment and lower change indicated less impairment.
Time Frame: Up to Month 24 of the core phase
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug in the core phase and had baseline and at least 1 post-dose primary efficacy measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: change in score per year
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1084 | 1062
change in score per year | 0.934 [0.838 to 1.030] | 0.926 [0.828 to 1.024]
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; Based on the linear mixed effects model, which included assessment time and treatment group by assessment time interaction as covariate with random intercept and slope; Test type: Superiority; p = 0.9088, Linear mixed effects model; Difference of Mean Slope = -0.008, 95% CI 2-sided [-0.145 to 0.129]

8. Secondary Outcome: Core Phase: Time to Worsening of CDR Score up to Month 24
Description: The CDR scale is a clinical global rating scale that requires interviewing both the participant and an informant who knows and has contact with the participant. The CDR scale is a clinician directed assessment of both cognition and function, and is intended to capture the state and therefore the disease stage of the participant. The CDR scale assesses 6 domains of participant function (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment=0, questionable impairment=0.5, mild impairment=1, moderate impairment=2 and severe impairment=3. The global CDR score is computed via an algorithm and ranges from 0 to 3. Higher score indicates more impairment. In this outcome measure, time (in months) to worsening of CDR score (that is, an increase from baseline by at least 0.5 points on the global CDR scale on 2 consecutive scheduled visits) up to month 24 was calculated.
Time Frame: Up to Month 24 of the core phase
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1084 | 1062
months | NA [NA to NA] — Median and 95 percent (%) confidence interval (CI) could not be estimated due to the low number of participants with events. | NA [24.07 to NA] — Median and Upper limit of 95% CI could not be estimated due to the low number of participants with events.
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; Based on a Cox regression model which included treatment group, clinical disease staging (MCI/Prodromal, mild AD), concurrent AD medication use, region, APOE4 status (positive, negative) as covariate; Test type: Superiority; p = 0.6155, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.77 to 1.16]

9. Secondary Outcome: Core Phase: Time to Conversion to Dementia for Participants Who Were Not Clinically Staged as Having Dementia at the Core Phase Baseline up to Month 24
Description: Time (in months) to conversion to dementia for participants who were not clinically staged as having dementia at the core phase baseline (that is time from randomization to conversion to dementia in clinical diagnosis).
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug in the core phase and had baseline and at least 1 post-dose primary efficacy measurement. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 902 | 901
months | 23.05 [21.14 to 24.66] | 21.40 [20.45 to 24.43]
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; Based on a Cox regression model which included treatment group, concurrent AD medication use, region, APOE4 status (positive, negative) as covariate; Test type: Superiority; p = 0.1281, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.96 to 1.35]

10. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the Alzheimer's Disease Assessment Scale-cognition14 (ADAS-Cog14) Score
Description: ADAS-cog14 is a psychometric instrument that evaluates 14-items (Immediate Word-recall [0-10], Commands [0-5], Constructional Praxis [0-5], Delayed Word-recall [0-10], Naming Objects/Fingers [0-5], Ideational Praxis [0-5], Orientation[0-8], Word Recognition [0-12], Remembering Test Instructions [0-5], Comprehension[0-5], Word Finding Difficulty [0-5], Spoken Language Ability [0-5], Executive Function [0-5], and Number Cancellation [0-5] test). It is considered to be more sensitive for less impaired populations such as MCI/Prodromal and mild AD participants. The total score ranges from 0 to 90. Higher score indicates more impairment.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1010 | 972
score on a scale | 5.38 (0.490) | 4.95 (0.520)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.525, MMRM; LS Mean Difference = -0.43, 95% CI 2-sided [-1.75 to 0.90]

11. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the MMSE Score
Description: The MMSE is a cognitive instrument commonly used for screening purposes, for staging of disease severity and is often measured longitudinally in AD clinical studies to follow disease progression and treatment effects. MMSE is composed of 30 questions grouped into domains (Orientation to Time [0-5], Orientation to Place [0-5], Registration [0-3], Attention and Calculation [0-5], Recall [0-3], Naming [0-2], Repetition [0-1], Comprehension [0-3], Reading [0-1], Writing [0-1], Drawing [0-1]). For each of the MMSE domains, six items are computed (Orientation to Time [0-5], Orientation to Place [0-5], Registration [0-3], Attention and Calculation [0-5], Recall [0-3], Language: Naming, Repetition, Comprehension, Reading, Writing, and Drawing [0-9]). The MMSE Total Score is the sum of the six domains and ranges from 0 to 30. If any domain score was missing then the total score was missing. Higher score indicates better function.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1056 | 1017
score on a scale | -2.87 (0.234) | -2.87 (0.241)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.977, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.64 to 0.62]

12. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the Functional Assessment Questionnaire (FAQ) Score
Description: FAQ scores 10 items & measures activities of daily living (paying bills/balancing checkbook, assembling tax records, shopping alone for clothes or groceries, playing game of skill such as bridge or chess/working on a hobby, heating water & turning off stove, preparing balanced meal, keeping track of current events, paying attention & understanding television program, remembering appointments, driving or traveling out of neighborhood). Each item is rated as follows: 0=Normal, 1=Has difficulty but does by self, 2=Requires assistance, 3=Dependent, or 8=Not Applicable. The total score is the sum of all 10 items & ranges from 0 to 30. Higher score indicates more impairment. If any activity was missed, then the total score was missed. Activities rated as "Not Applicable" were not used in the computation of the total score. To account for "Not Applicable" activity, the total score was weighted as:Total Score=Total Score*30/(30 minus 3 times the number of activities marked"Not Applicable").
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1038 | 1001
score on a scale | 5.20 (0.448) | 5.32 (0.459)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.854, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-1.09 to 1.32]

13. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the ADAS-cog14 Word List (Immediate Recall and Delayed Recall) Score
Description: The ADAS-cog14 Word List is a summation of two items: "Immediate Word-recall" and "Delayed Word-recall". Immediate Word-recall test: Participants are asked to recall words and the number of "No" responses for each trial (total 3 trials) are summed. Subscore: sum of scores from 3 trials, divided by 3. Score ranges from 0 to 10. Delayed Word-recall: Participants used to recall words after a delay and the number of "No" responses are summed. Score ranges from 0 to 10. The Total Score ranges from 0 to 20. Higher score indicates more impairment.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1050 | 1005
score on a scale | 1.63 (0.195) | 1.36 (0.207)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.314, MMRM; LS Mean Difference = -0.27, 95% CI 2-sided [-0.79 to 0.26]

14. Secondary Outcome: Core Phase: Change From Baseline up to Month 24 in the Alzheimer's Disease Assessment Scale-cognition11 (ADAS-Cog11) Score
Description: ADAS-cog11 is a psychometric instrument that evaluates 11-items (Immediate Word-recall [0 to 10], Commands [0-5], Constructional Praxis [0-5], Naming Objects/Fingers [0-5], Ideational Praxis [0-5], Orientation[0-8], Word Recognition [0-12], Remembering Test Instructions [0-5], Comprehension[0-5], Word Finding Difficulty [0-5], Spoken Language Ability [0-5] test) and is considered more sensitive for less impaired populations such as MCI/Prodromal and mild AD participants. The Total score ranges from 0 to 70. Higher score indicates more impairment.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 24 of the core phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 1010 | 972
score on a scale | 4.11 (0.370) | 4.18 (0.391)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.895, MMRM; LS Mean Difference = 0.07, 95% CI 2-sided [-0.93 to 1.07]

15. Secondary Outcome: Core Phase: Change From Last Dose in the CDR-SB Score
Description: The CDR scale is a clinical global rating scale that requires interviewing both the participant and an informant who knows and has contact with the participant. The CDR scale is a clinician directed assessment of both cognition and function, and is intended to capture the state and therefore the disease stage of the participant. The CDR scale assesses 6 domains of participant function (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment=0, questionable impairment=0.5, mild impairment=1, moderate impairment=2 and severe impairment=3. The CDR-SB is a sum of the individual domain scores and ranges from 0 to 18. Higher score indicates more impairment.
Time Frame: From last dose in the core phase (up to Month 24) up to 3 months follow up (up to Month 27)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 759 | 734
score on a scale | 0.40 (0.045) | 0.44 (0.046)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; Analysis was based on the MMRM and factors for treatment group, visit, treatment group by visit interaction, clinical disease staging (MCI/Prodromal, mild AD), concurrent AD medication use, region, ApoE4 status (positive, negative) as fixed effects, and the baseline value as covariate; Test type: Superiority; p = 0.542, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.09 to 0.17]

16. Secondary Outcome: Core Phase: Change From Last Dose in the ADCOMS
Description: ADCOMS is a weighted linear combination of 12 items from three existing clinical scales: the ADAS-cog, the MMSE, and the CDR. Four items are from the ADAS-cog (A4 [Delayed Word Recall], A7 [Orientation], A8 [Word Recognition], A11 [Word Finding]); 2 items are from the MMSE (M1 [Orientation Time], M7 [Drawing]); 6 items are from the CDR (C1 [Personal Care], C2 [Community Affairs], C3 [Home and Hobbies], C4 [Judgment and Problem Solving], C5 [Memory], C6 [Orientation]). Composite score is derived from the variables from the 12 items, and ranges from 0 to 1.97, where higher score indicates worse performance.
Time Frame: From last dose in the core phase (up to Month 24) up to 3 months follow-up (up to Month 27)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 666 | 646
score on a scale | 0.06 (0.005) | 0.06 (0.005)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.380, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.02 to 0.01]

17. Secondary Outcome: Core Phase: Change From Last Dose in the ADAS-cog11 Score
Description: as for outcome 14
Time Frame: From last dose in the core phase (up to Month 24) up to 3 months follow-up (up to Month 27)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 679 | 647
score on a scale | 0.95 (0.150) | 0.56 (0.153)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.063, MMRM; LS Mean Difference = -0.40, 95% CI 2-sided [-0.82 to 0.02]

18. Secondary Outcome: Core Phase: Change From Last Dose in the ADAS-cog14 Score
Description: ADAS-cog14 is a psychometric instrument that evaluates 14-items (Immediate Word-recall [0 to 10], Commands [0-5], Constructional Praxis [0-5], Delayed Word-recall [0-10], Naming Objects/Fingers [0-5], Ideational Praxis [0-5], Orientation[0-8], Word Recognition [0-12], Remembering Test Instructions [0-5], Comprehension[0-5], Word Finding Difficulty [0-5], Spoken Language Ability [0-5], Executive Function [0-5], and Number Cancellation [0-5] test). It is considered to be more sensitive for less impaired populations such as MCI/Prodromal and mild AD participants. The Total Score ranges from 0 to 90. Higher score indicates more impairment.
Time Frame: From last dose in the core phase (up to Month 24) up to 3 months follow-up (up to Month 27)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 679 | 647
score on a scale | 0.96 (0.196) | 0.40 (0.201)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.045, MMRM; LS Mean Difference = -0.56, 95% CI 2-sided [-1.11 to -0.01]

19. Secondary Outcome: Core Phase: Change From Last Dose in the MMSE Score
Description: as for outcome 11
Time Frame: From last dose in the core phase (up to Month 24) up to 3 months follow-up (up to Month 27)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 734 | 719
score on a scale | -0.22 (0.101) | -0.26 (0.102)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.799, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.32 to 0.24]

20. Secondary Outcome: Core Phase: Change From Last Dose in the ADAS-cog14 Word List (Immediate Recall and Delayed Recall) Score
Description: as for outcome 13
Time Frame: From last dose in the core phase (up to Month 24) up to 3 months follow-up (up to Month 27)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 707 | 685
score on a scale | 0.54 (0.088) | 0.22 (0.090)
Statistical Analysis 1: Comparison: Core Phase: Placebo vs Core Phase: Elenbecestat 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.012, MMRM; LS Mean Difference = -0.32, 95% CI 2-sided [-0.56 to -0.07]

21. Secondary Outcome: Extension Phase: Change From Core Phase Baseline up to Month 12 of the Extension Phase in CDR-SB Score
Description: as for outcome 15
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: Data could not be reported as the study was terminated prior to reaching the specified time point for assessment in the extension phase. Statistical analysis plan was modified to indicate that the extension phase analysis was not done.
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

22. Secondary Outcome: Extension Phase: Change From Core Phase Baseline up to Month 12 of the Extension Phase in ADCOMS
Description: as for outcome 16
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: as for outcome 21
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

23. Secondary Outcome: Extension Phase: Change From Core Phase Baseline up to Month 12 of the Extension Phase in MMSE Score
Description: The MMSE is a cognitive instrument commonly used for screening purposes, for staging of disease severity and is often measured longitudinally in AD clinical studies to follow disease progression and treatment effects. MMSE is composed of 30 questions grouped into domains (Orientation to Time [0-5], Orientation to Place [0-5], Registration [0-3], Attention and Calculation [0-5], Recall [0-3], Naming [0-2], Repetition [0-1], Comprehension [0-3], Reading [0-1], Writing [0-1], Drawing [0-1]). For each of the MMSE domains, six items are computed (Orientation to Time [0-5], Orientation to Place [0-5], Registration [0-3], Attention and Calculation [0-5], Recall [0-3], Language: Naming, Repetition, Comprehension, Reading, Writing, and Drawing [0-9]). The MMSE Total Score is the sum of the six domains and ranges from 0 to 30. If any domain score is missing then the total score is missing. Higher score indicates better function.
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: as for outcome 21
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

24. Secondary Outcome: Extension Phase: Change From Core Phase Baseline up to Month 12 of the Extension Phase in FAQ Score
Description: as for outcome 12
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: as for outcome 21
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

25. Secondary Outcome: Extension Phase: Change From Core Phase Baseline up to Month 12 of the Extension Phase in ADAS-cog14 Score
Description: as for outcome 18
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: as for outcome 21
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

26. Secondary Outcome: Extension Phase: Change From Core Phase Baseline up to Month 12 of the Extension Phase in ADAS-cog14 Word List (Immediate Recall and Delayed Recall) Score
Description: as for outcome 13
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: as for outcome 21
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

27. Secondary Outcome: Extension Phase: Time to Conversion to Dementia for Participants Who Were Not Clinically Staged as Having Dementia at the Core Phase Baseline up to Month 12 of the Extension Phase
Description: as for outcome 9
Time Frame: Baseline (Day 1: before first dose in the core phase) up to Month 12 of the extension phase
Population: as for outcome 21
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 27 months (including 3 months follow up) for the Core Phase and up to approximately 6 months (including 1 month follow up) for the Extension Phase
Description: In the Core Phase, adverse events were reported for the SAS (the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment). In the Extension Phase, adverse events were reported for the All Safety Participants analysis set: the group of participants who enrolled into the extension phase and received at least 1 dose of study drug in the extension phase.
Groups:
- Extension Phase: Elenbecestat 50 mg: Eligible participants who completed the core phase entered the extension phase and received one elenbecestat 50 mg tablet, orally, once daily in the morning with or without food until commercial availability of elenbecestat, or a lack of positive benefit-risk assessment was determined, whichever occurred first. Participants were followed up for 1 month after last dose of elenbecestat in extension phase.
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 50 mg | Extension Phase: Elenbecestat 50 mg
All-Cause Mortality (participants affected / at risk) | 6/1105 | 3/1099 | 0/18
Serious Adverse Events (participants affected / at risk) | 117/1105 | 134/1099 | 0/18
Other Adverse Events (participants affected / at risk) | 292/1105 | 391/1099 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Placebo (N=1105) | Core Phase: Elenbecestat 50 mg (N=1099) | Extension Phase: Elenbecestat 50 mg (N=18)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 4 (5) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 3 (4) | 0 (0)
Idiopathic orbital inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Placebo (N=1105) | Core Phase: Elenbecestat 50 mg (N=1099) | Extension Phase: Elenbecestat 50 mg (N=18)
Lymphopenia (Blood and lymphatic system disorders) | 18 (18) | 70 (89) | 0 (0)
Nasopharyngitis (Infections and infestations) | 67 (80) | 71 (86) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 50 (56) | 58 (63) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 55 (79) | 66 (101) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 60 (71) | 61 (79) | 0 (0)
Dizziness (Nervous system disorders) | 45 (49) | 57 (61) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 36 (42) | 57 (66) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 22 (26) | 60 (78) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to an unfavorable risk-benefit ratio including no evidence of potential efficacy and the adverse event profile in participants with drug treatment was worse than that in participants who received placebo. The small sample size at the 24 month time point of the core phase limits the interpretability of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT02956486/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT02956486/SAP_001.pdf